CLINICAL TRIAL: NCT00876382
Title: Community Oncology Setting Disease Outcomes of Sorafenib (Nexavar) Use in Advanced Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: SCRI OUTCOMES 06
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Renal Cell Carcinoma
Keywords: advanced renal cell carcinoma; renal cancer; renal cell; Sorafenib; Nexavar; Bevacizumab; Avastin; Sunitinib; Sutent
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A retrospective medical record abstraction study of at least 200 advanced renal cell carcinoma patients treated in the following settings:

* Patients with advanced renal cell carcinoma treated with Sorafenib (Nexavar) as second-line therapy after Sunitinib (Sutent) or Bevacizumab (Avastin) for first-line therapy (about 100 patients)
* Patients with advanced renal cell carcinoma treated with Sorafenib (Nexavar) as first-line therapy followed by Sunitinib (Sutent) as second-line therapy (about 100 patients)

DETAILED DESCRIPTION:
Recently, a number of targeted agents have demonstrated single-agent activity in the treatment of advanced renal cell carcinoma. Bevacizumab, a humanized monoclonal antibody directed against VEGF, resulted in an improvement in median progression-free survival when compared to placebo in a prospective, randomized trial. More recently, the multitargeted agents sorafenib and sunitinib have been approved for use in the treatment of advanced renal cell carcinoma. Both have proven superior to previous interferon and other standard treatment; however it is not clear how these drugs should be used in the treatment sequence. With roughly 80% of cancer patients receiving their oncology care in the community setting, we are proposing a review and evaluation of at least 200 advanced renal cell carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patient cases are those that have received Sorafenib (Nexavar) as second-line therapy after Sunitinib (Sutent) or Bevacizumab (Avastin) for first-line therapy or those patients that were treated with Sorafenib (Nexavar) as first-line therapy followed by Sunitinib (Sutent) as secondline therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two hundred plus patients treated with Nexavar as first or second line therapy for advanced renal cell carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2009-05; Primary Completion 2011-02 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of Nexavar as second-line therapy in patients with advanced renal cell carcinoma treated with Nexavar after first-line therapy with Sutent or Avastin. | 6 months

SECONDARY OUTCOMES:
To evaluate safety and efficacy of Nexavar as first-line therapy in patients with advanced renal cell carcinoma and as first-line therapy followed by Sutent as second-line therapy in patients with advanced renal cell carcinoma. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Patton, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (8):
- United States (8):
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - Gulfcoast Oncology Associates, St. Petersburg, Florida
  - Medical Oncology Associates of Augusta, Augusta, Georgia
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Jackson Oncology Associates, Jackson, Mississippi
  - St. Louis Cancer Care, Chesterfield, Missouri
  - Oncology Hematology Care, Cincinnati, Ohio
  - Tennessee Oncology, PLLC, Nashville, Tennessee